CLINICAL TRIAL: NCT04266405
Title: Efficacy Testing of Collagen and Zhuyin Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20-003-B
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- Collagen and Zhuyin Drinks (Experimental)
  Interventions: Dietary Supplement: Collagen Cubilose Drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 1 bottle (50 mL) per day for 28 days
  Arms: Placebo drink
Dietary Supplement: Collagen Cubilose Drink — consume 1 bottle (50 mL) per day for 28 days
  Arms: Collagen and Zhuyin Drinks

SUMMARY:
To assess collagen and zhuyin drink on skin & body condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, heart, liver, kidney, endocrine and other organs and patients with mental illness (according to medical history).
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure in the past 4 weeks.
* Vegetarian
* Subjects who have large spots (area >3 square centimeter) or abnormal acne.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The change of skin moisture | Change from Baseline skin moisture at 4 weeks
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin wrinkles | Change from Baseline skin wrinkles at 4 weeks
  VISIA Complexion Analysis System was utilized to measure wrinkles. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 4 weeks
  DermaLab® USB - 20 MHz High Freq. Ultrasound probe was utilized to scan and analyze skin collagen density. Units:Intensity score
The change of TEWL | Change from Baseline TEWL at 4 weeks
  Tewameter® TM 300 was utilized to measure TEWL. Units: g/h/m2
The change of skin brightness | Change from Baseline skin brightness at 4 weeks
  Glossymeter GL 200 was utilized to measure skin brightness. Units: arbitrary units
The change of interleukin-6 | Change from Baseline skin brightness at 4 weeks
  Venous blood was sampled to measure concentrations of interleukin-6.
The change of interleukin-8 | Change from Baseline skin brightness at 4 weeks
  Venous blood was sampled to measure concentrations of interleukin-8.
The change of Tumor necrosis factor | Change from Baseline skin brightness at 4 weeks
  Venous blood was sampled to measure concentrations of Tumor necrosis factor.
The change of Matrix metalloproteinase-1 | Change from Baseline skin brightness at 4 weeks
  Venous blood was sampled to measure concentrations of Matrix metalloproteinase-1 .
The change of metallopeptidase inhibitor 1 | Change from Baseline skin brightness at 4 weeks
  Venous blood was sampled to measure concentrations of metallopeptidase inhibitor 1.

SECONDARY OUTCOMES:
The change of skin texture | Change from Baseline skin texture at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin pores | Change from Baseline skin pores at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units
The change of skin spots | Change from Baseline skin spots at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin spots. Units: arbitrary units
The change of red areas | Change from Baseline red areas at 4 weeks
  VISIA Complexion Analysis System was utilized to measure red areas. Units: arbitrary units

CONTACTS AND LOCATIONS:
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan